CLINICAL TRIAL: NCT04089124
Title: Randomized Controlled Trial to Compare the Outcomes Of Zone II Flexor Tendon Repair of the Hand Under General Anesthesia Versus Wide Awake Local Anesthesia No Tourniquet
Brief Title: Compare the Outcomes of Zone II Flexor Tendon Repair of the Hand Under General Anesthesia Versus WALANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina S. Fekry, Demonstrator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zone II flexor repair
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cut Flexor Hand; Walant; General Anesthesia

STUDY DESIGN:
Intervention Model Description: repair zone II cut flexor of hand under GA and Walant
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repair using General anesthesia ( control group) (Other): Surgery repair zone II under GA
  Interventions: Procedure: surgery of zone II cut flexor repair
- repair using Walant (Other): Surgery repair zone II under WALANT
  Interventions: Procedure: surgery of zone II cut flexor repair

INTERVENTIONS:
Procedure: surgery of zone II cut flexor repair — we will repair tendon of FDP only using 6 strand technique using PDS 4/0 core suture - prolene 6/0 running suture

SUMMARY:
Comparison between results of repair of cut flexor zone II under General anesthesia and Walant

DETAILED DESCRIPTION:
Cut Flexor is common injury ,has unique characters as they cannot heal without surgical treatment, unique anatomy of the tendons running through flexor tendon sheaths to function and postoperative management &mobilization to prevent adhesions and improve gliding but risk of rupture.

The hand is divided into five zones (Verdan's). Zone II is described by Bunnel as "No Man's Land" historically back to 14th century (area outside London used for executions) because it was previously believed that primary repair should not be done in this zone. After understanding of flexor tendon anatomy, biomechanics , and healing new techniques of surgery and anesthesia repair is possible with good results.

General anesthesia has been the standard technique for along time. wide awake local anesthesia no tourniquet. (WALANT),using safe drugs lidocaine for anesthesia and epinephrine for hemostasis, the investigators can do operations while patient is awake.

WALANT has been recommended by some surgeons to be the next standard for repair of zone 2 injuries .

This techniques has a lot of Advantages in repair zone II as 1) intraoperative testing of the flexor repair by active movement to exclude any gap. and lets the surgeon see that the repair fits through the pulleys with active movement.

2)sheath and pulley damage are minimized, as flexor tendons are repaired through small transverse sheathotomy incisions 3) the surgeon can interview the patient during the procedure and assess the ability to comply with the postoperative regimen 4) the risks of general anesthesia are avoided in most patients. Negative effects of general anesthesia include nausea and vomiting, hospital admission for anesthesia recovery, exacerbation of comorbidity issues such as diabetes, aggressive flexion by the patient emerging from general anesthesia,and others

ELIGIBILITY:
Inclusion Criteria:

* Acute zone II flexor tendon injuries of the hand in both genders in medial four fingers.
* Cooperative patients aged between 16-60 years.
* Sharp mechanism of injury
* Single level injury

Exclusion Criteria:

* Age less than sixteen years old or more than sixty years old .
* Associated fractures close to the tendon injury.
* Vascular injury requiring revascularization
* Multiple level injury
* Combined flexor and extensor laceration
* Insufficient skin and soft tissue coverage
* Tendon substance loss

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
range of motions using Jamar finger goniometer | baseline (2 weeks, 1.5 months , 3 months , 4.5 months and 6 months .)
  The functions of treated fingers were calculated using original Strickland and Glogovac criteria

SECONDARY OUTCOMES:
complications | baseline
  as adhesion formation, which limits active range of motion. joint contracture, tendon rupture, triggering, and pulley failure with tendon bowstringin Infection or neuroma
Healing vs failure of repair | baseline
  if can move and use flexor tendons again or not
DASH score using DASH questionnaire | 6 months
  Disabilites of the Arm , Shoulder , Hand

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Wolfe SW, Pederson WC, Hotchkiss RN, Kozin SH , Cohen MS. Green's Operative Hand Surgery E-book. Elsevier Health sciences ; 2016 Feb 24.
- [Background] Canale ST, Beaty JH, Campbell WC. Campbell's operative orthopaedics. 2013.
- [Background] Lalonde D. Wide Awake Hand Surgery . CRC press. 2016 Jan 27.
- [Background] Griffin M, Hindocha S, Jordan D, Saleh M, Khan W. An overview of the management of flexor tendon injuries. Open Orthop J. 2012;6:28-35. doi: 10.2174/1874325001206010028. Epub 2012 Feb 23. PMID 22431948
- [Background] Farnebo S, Chang J. Practical management of tendon disorders in the hand. Plast Reconstr Surg. 2013 Nov;132(5):841e-853e. doi: 10.1097/PRS.0b013e3182a48ccf. PMID 24165636
- [Background] Steiner MM, Calandruccio JH. Use of Wide-awake Local Anesthesia No Tourniquet in Hand and Wrist Surgery. Orthop Clin North Am. 2018 Jan;49(1):63-68. doi: 10.1016/j.ocl.2017.08.008. PMID 29145985
- [Background] Pires Neto PJ, Moreira LA, Las Casas PP. Is it safe to use local anesthesia with adrenaline in hand surgery? WALANT technique. Rev Bras Ortop. 2017 Jul 19;52(4):383-389. doi: 10.1016/j.rboe.2017.05.006. eCollection 2017 Jun-Jul. PMID 28884094
- [Background] Lalonde DH, Kozin S. Tendon disorders of the hand. Plast Reconstr Surg. 2011 Jul;128(1):1e-14e. doi: 10.1097/PRS.0b013e3182174593. PMID 21701291
- [Background] Lalonde DH. Latest Advances in Wide Awake Hand Surgery. Hand Clin. 2019 Feb;35(1):1-6. doi: 10.1016/j.hcl.2018.08.002. PMID 30470325
- [Background] Higgins A, Lalonde DH, Bell M, McKee D, Lalonde JF. Avoiding flexor tendon repair rupture with intraoperative total active movement examination. Plast Reconstr Surg. 2010 Sep;126(3):941-945. doi: 10.1097/PRS.0b013e3181e60489. PMID 20463621
- [Background] Festen-Schrier VJMM, Amadio PC. Wide Awake Surgery as an Opportunity to Enhance Clinical Research. Hand Clin. 2019 Feb;35(1):93-96. doi: 10.1016/j.hcl.2018.08.003. PMID 30470336
- [Background] Osada D, Fujita S, Tamai K, Yamaguchi T, Iwamoto A, Saotome K. Flexor tendon repair in zone II with 6-strand techniques and early active mobilization. J Hand Surg Am. 2006 Jul-Aug;31(6):987-92. doi: 10.1016/j.jhsa.2006.03.012. PMID 16843161
- [Background] Wong YR, Lee CS, Loke AM, Liu X, Suzana MJ I, Tay SC. Comparison of Flexor Tendon Repair Between 6-Strand Lim-Tsai With 4-Strand Cruciate and Becker Technique. J Hand Surg Am. 2015 Sep;40(9):1806-11. doi: 10.1016/j.jhsa.2015.05.007. Epub 2015 Jun 30. PMID 26142080
- [Background] Kleinert HE, Spokevicius S, Papas NH. History of flexor tendon repair. J Hand Surg Am. 1995 May;20(3 Pt 2):S46-52. doi: 10.1016/s0363-5023(95)80169-3. No abstract available. PMID 7642949